CLINICAL TRIAL: NCT07266792
Title: An Open Label, Randomized, Two-period, Twotreatment, Two-sequence, Truncated, Crossover, Balanced, Single Dose Oral Bioequivalence Study.
Brief Title: Bioequivalence Study to Compare Brexpiprazole 4 mg Film Coated Tablets Versus RXULTI 4 mg Film Coated Tablet (Brexpiprazole)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: C1B05603
Record Dates: First submitted 2025-12-04; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brexpiprazole Film Coated Tablets (Experimental): Brexpiprazole 4 mg Film Coated Tablets
  Interventions: Drug: Brexpiprazole Film Coated Tablets; Drug: RXULTI film coated tablet
- RXULTI film coated tablet (Active Comparator): RXULTI 4 mg film coated tablet (Brexpiprazole)
  Interventions: Drug: Brexpiprazole Film Coated Tablets; Drug: RXULTI film coated tablet

INTERVENTIONS:
Drug: Brexpiprazole Film Coated Tablets — 1 tablet of Brexpiprazole 4 mg Film Coated Tablets
Drug: RXULTI film coated tablet — 1 tablet of RXULTI 4 mg film coated tablet (Brexpiprazole)

SUMMARY:
Single dose oral bioequivalence study of Brexpiprazole 4 mg Film Coated Tablets and RXULTI® (Brexpiprazole) 4 mg film-coated tablets in healthy adult human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Age: 45 to 65 years old, both inclusive.
* Gender: Male and/or non-pregnant, non-lactating female.
* A. Female of child-bearing potential had a negative serum beta human chorionic gonadotropin (β-HCG) pregnancy test performed within 28 days of the first dose of study medication. They must use an acceptable form of contraception. For female of child-bearing potential, acceptable forms of contraception included the following:
* i. Non hormonal intrauterine device in place for at least 3 months prior to the start of the study and remaining in place during the study period, or
* ii. Barrier methods containing or used in conjunction with a spermicidal agent, or
* iii. Surgical sterilization or
* iv. Practicing sexual abstinence throughout the course of the study.
* B. Female were not considered of child-bearing potential if one of the following was reported and documented on the medical history:
* i. Postmenopausal with spontaneous amenorrhea for at least one year, or
* ii. Spontaneous amenorrhea for more than 6 months and less than one year with Serum Follicular Stimulating Hormone (FSH) level > 40 mIU/mL, or
* iii. Bilateral oophorectomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or
* iv. Total hysterectomy and an absence of bleeding for at least 3 months.
* 3) BMI: 18.5 to 30.0 kg/m2, both inclusive; BMI value should be rounded off to one significant digit after decimal point (e.g. 30.04 rounds down to 30.0, while 18.45 rounds up to 18.5).
* 4) Non-smokers and non-tobacco user (i.e. had no past history of smoking and tobacco consumed for at least one year prior to study).
* 5) Was able to communicate effectively with study personnel.
* 6) Was willing to provide written informed consent to participate in the study.
* 7) All volunteers were judged by the principal or sub-investigator or physician as normal and healthy during a pre-study safety assessment performed within 28 days of the first dose of study medication which included:
* a) A physical examination (clinical examination) with no clinically significant finding.
* No additional tests and/or examinations were performed.
* All results were assessed against the current laboratory normal ranges at the time of testing and a copy of the normal ranges used was included in the study documentation.

Exclusion Criteria:

* 1) Had history of allergic responses to Brexpiprazole or other related drugs, or any of its formulation ingredients.
* 2) Had significant diseases or clinically significant abnormal findings during screening [medical history, physical examination (clinical examination), laboratory evaluations, ECG recording, gynecological history and examination (including pelvic examination and routine breast examination) (for female volunteers)].
* 3) Any disease or condition like diabetes, psychosis or others, which might compromise the haemopoietic, gastrointestinal, renal, hepatic, cardiovascular, respiratory, Central nervous system or any other body system.
* 4) Had history or presence of bronchial asthma.
* 5) Used any hormone replacement therapy within 3 months prior to the first dose of study medication.
* 6) Used any depot injection or implant of any drug within 3 months prior to the first dose of study medication.
* 7) Used CYP enzyme inhibitors or inducers within 30 days prior to the first dose of study medication (see https://drug-interactions.medicine.iu.edu/MainTable.aspx).
* 8) Had history or evidence of drug dependence or of alcoholism or of moderate alcohol use.
* 9) Had history of difficulty with donating blood or difficulty in accessibility of veins.
* 10) A positive hepatitis screen (includes subtypes B & C).
* 11) A positive test result for HIV antibody.
* 12) Volunteer who had received a known investigational drug within seven elimination half-life of the administered drug prior to the first dose of study medication.
* 13) Volunteer who had donated blood or loss of blood 50 ml to 100 ml within 30 days or 101 ml to 200 ml within 60 days or >200 ml within 90 days (excluding volume drawn at screening for this study) prior to first dose of study medication, whichever was greater.
* 14)Had history of difficulty in swallowing or of any gastrointestinal disease, which could affect drug absorption.
* 15) Intolerance to venipuncture
* 16) Any food allergy, intolerance, restriction or special diet that, in the opinion of the principal investigator or sub-investigator, could contraindicate the volunteer's participation in this study.
* 17) Institutionalized volunteer.
* 18) Used any prescribed medications within 14 days prior to the first dose of study medication.
* 19) Used any OTC products, vitamin and herbal products, etc., within 7 days prior to the first dose of study medication.
* 20) Used grapefruit and grapefruit containing products within 7 days prior to the first dose of study medication.
* 21) Ingestion of any caffeine or xanthine products (i.e. coffee, tea, chocolate, and caffeine-containing sodas, colas, etc.), recreational drugs, alcohol or other alcohol containing products within 48 hours prior to the first dose of study medication.
* 22) Ingestion of any unusual diet, for whatever reason (e.g.: low sodium) for three weeks prior to the first dose of study medication.
* 23) Volunteer with WBC and neutrophil count less than lower limit of normal range.
* 24) Volunteers with history of Psychosis, Suicidal thoughts and behavior or Stroke, Transient ischemic attack (TIA), Seizure or any other related medical condition.
* 25) Volunteers with QTc interval more than 450 ms on ECG measurement at the time of screening.
* 26) Sitting systolic blood pressure less than 110 mmHg or greater than 140 mmHg or sitting diastolic blood pressure less than 70 mmHg or greater than 90 mmHg and pulse rate less than 60 or greater than 100 beats per minute during screening.
* 27) Volunteer had a personal or family history of dystonic reactions to medications.
* 28)Had history of use of any neuroleptic drugs and illicit drugs.
* 29)Had history of Hyperglycemia.
* 30)Had history of Myocardial Infarction/ Ischaemic heart disease.
* 31)Had history of Venous Thromboembolism.
* 32)Had history of a known history of Extrapyramidal Symptoms (EPS).
* 33)Had history of Dementia and Tardive Dyskinesia.
* 34)Had history of Dysphagia.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2025-06-22 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Maximum measured plasma concentration over the time span specified (Cmax) | 72 hours
  The 90% confidence interval of the relative mean (Geometric least square mean) of test to reference product for Ln-transformed Pharmacokinetic parameters Cmax
Area under the plasma concentration-time curve from time point to the 72 hours (AUC72) | 72 hours
  The 90% confidence interval of the relative mean (Geometric least square mean) of test to reference product for Ln-transformed Pharmacokinetic parameters AUC72

SECONDARY OUTCOMES:
Time of the maximum measured plasma concentration (Tmax) | 72 hours
  Descriptive Statistics

CONTACTS AND LOCATIONS:
Locations (1):
- Cliantha Research Limited, Ahmedabad, Gujarat, India